CLINICAL TRIAL: NCT01717547
Title: Strength and Awareness in Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Brenner, Director, VA Eastern Colorado Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0641
Record Dates: First submitted 2012-08-29; First posted 2012-10-30 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Stress Disorders
Keywords: Veterans; Yoga; Stress
MeSH Terms: conditions — Stress Disorders, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga (Experimental): Yoga-based treatment - manualized group treatment - classes will be held twice per week for approximately 85 minutes for a period of eight weeks.
  Interventions: Behavioral: Yoga-based treatment

INTERVENTIONS:
Behavioral: Yoga-based treatment

SUMMARY:
The aims of this research study are to 1) assess the acceptability and feasibility of conducting a yoga-based intervention for Veterans receiving care at a Veterans Affairs Medical Center, and 2) obtain preliminary data regarding the effect of the intervention on Veteran's mental health.

DETAILED DESCRIPTION:
Since October of 2001, approximately over 2 million troops have been deployed in the Global War on Terror. Many service members are returning with both physical injuries and mental health conditions. High rates of both post traumatic stress disorder (PTSD) and/or mild traumatic brain injury (mTBI) and associated symptoms have been noted. It has been estimated that approximately 18-20% of returning service members meet criteria for PTSD and that 11-23% of veterans have a history of mTBI. It has been well established in the research literature that these two conditions frequently co-occur. While there is a dearth of evidence-based treatment for co-occurring PTSD and mTBI, it has been suggested that best practices entail treating presenting symptoms (hyperarousal, hypo-arousal, emotional reactivity, irritability, depression, anxiety, concentration problems) regardless of etiology. Yoga may be particularly well-suited to treating returning servicemen as data suggests that core symptoms that develop with a history of trauma exposure (e.g: hyperarousal; hypoarousal; emotional reactivity; anxiety, irritability), are physiologically based, somatically experienced and often not amenable to change through talking alone. In addition, yoga may assist with dysregulation often associated with mental health and physical conditions, and facilitate the development of mindfulness skills. Research suggests that that moment-to-moment awareness of present experience may decrease emotional reactivity and anxiety, and increase the capacity for self-regulation. Mindfulness skills have also been associated with: building resilience in the midst of stress; allowing one to better cope with physical discomfort; decreasing anxiety and depression; decreasing reactivity. All of these areas are relevant to improving the health and well-being of Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veterans receiving care by a primary care provider at DVAMC
* Between the ages of 18 and 50
* Able to provide informed consent
* Able to adequately answer comprehension questions
* Documented VA primary care provider medical clearance to participate in the study as noted on the medical clearance form

Exclusion Criteria:

* Veterans younger than 18, or older than 50 years of age
* Inability to provide informed consent
* Inability to answer comprehension questions
* Meet criteria for active substance dependence, excluding Cannabis dependence as determined by clinical interview
* Identification of active psychosis as determined by clinical interview
* Documentation on the medical clearance form by VA primary care provider which suggests barriers to Veteran participation
* Veterans whom have sustained an amputation and/or whom have limited physical mobility as documented by the VA primary care provider
* Veterans already participating in an ongoing yoga practice of up to two times weekly

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Distress | Change from baseline to approximately 8 weeks
  Change in OQ 45 Scores pre and post intervention

SECONDARY OUTCOMES:
Change in Acceptability | Change in baseline up to 8 weeks post
  To assess participant satisfaction post-intervention using the Client Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brenner, PhD, Principal Investigator — VA ECHCS
Locations (1):
- Denver Veterans Affairs Medical Center, Denver, Colorado, United States

REFERENCES:
- See also: VA VISN 19 MIRECC website — http://www.mirecc.va.gov/visn19/